CLINICAL TRIAL: NCT01326546
Title: A Randomized, Double-blind, Multicenter Phase II Clinical Trial to Evaluate the Efficacy and Safety of Therapeutic Hepatitis B Vaccine (Mimogen-based) Joint Entecavir in Treating HBeAg Positive Chronic Hepatitis B Patients
Brief Title: Therapeutic Hepatitis B Vaccine (Mimogen-based) Joint Entecavir in Treating Chronic Hepatitis B Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chongqing Jiachen Biotechnology Ltd. (Industry)
Collaborators: Third Military Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 71006.04
Record Dates: First submitted 2011-03-28; First posted 2011-03-31 (Estimated); Results first posted 2019-06-26 (Actual); Last update posted 2019-06-26 (Actual); Status verified 2019-03

CONDITIONS: Chronic Hepatitis B
Keywords: Therapeutic HBV Vaccine; Chronic Hepatitis B; HBeAg positive; HBV-specific Cytotoxic T Lymphocyte
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — entecavir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Therapeutic HBV vaccine+Entecavir (Experimental): Inject εPA-44 900μg at week 0, 3, 6, 9, 12, 15, 18, 21, 24, 28, 32, 36, 40, 44, 48 and Oral intake entecavir 0.5mg per day.
  Interventions: Biological: Therapeutic HBV vaccine; Drug: entecavir
- placebo+Entecavir (Placebo Comparator): Placebo comparator: Inject placebo 900μg at week 0, 3, 6, 9, 12, 15, 18, 21, 24, 28, 32, 36, 40, 44, 48 and Oral intake entecavir 0.5mg per day.
  Interventions: Drug: entecavir; Other: placebo

INTERVENTIONS:
Biological: Therapeutic HBV vaccine — Inject εPA-44 900μg at week 0, 3, 6, 9, 12, 15, 18, 21, 24, 28, 32, 36, 40, 44, 48.
  Other Names: εPA-44
  Arms: Therapeutic HBV vaccine+Entecavir
Drug: entecavir — 0.5mg,per day,oral intake.
  Other Names: Baraclude
Other: placebo — Inject placebo 900μg at week 0, 3, 6, 9, 12, 15, 18, 21, 24, 28, 32, 36, 40, 44, 48.
  Other Names: empty liposome
  Arms: placebo+Entecavir

SUMMARY:
The purpose is to evaluate efficacy and safety of therapeutic hepatitis B virus (HBV) vaccine (mimogen-based)) Joint entecavir treatment in chronic hepatitis B patients.

DETAILED DESCRIPTION:
Eligible subjects are enrolled and assigned into 2 groups randomly with a 1:1 ratio：

1. Therapeutic HBV vaccine Joint Entecavir group：Inject εPA-44 900μg at week 0, 3, 6, 9, 12, 15, 18, 21, 24, 28, 32, 36, 40, 44, 48 + Oral intake entecavir 0.5mg per day ；
2. Empty liposome Joint Entecavir group：Inject empty liposome at week 0, 3, 6, 9, 12, 15, 18, 21, 24, 28, 32, 36, 40, 44, 48 + Oral intake entecavir 0.5mg per day.

The study cycle consists of screening and enrollment period (week -4～0), treatment and follow-up period (week 0-96).

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-65 years, male or female;
2. Conforming to diagnosis standard of chronic hepatitis B according to " 2005 Guideline for Prevention and Treatment of Hepatitis B " , (with positive HBsAg for more than 6 months), never have systemic treatment of anti-HBV viral ,and

   * HBV-DNA ≥ 1.72×10^4 IU/ml；
   * HBeAg (+), HBeAb (-)；
   * ALT within 2 to 10 times of ULN (upper limits of normal);
3. HLA-A2 positive;
4. Compensatory liver disease having following hematological and biochemical parameters:

   * WBC ≥ 3.5×10^9/L;
   * ANC ≥ 1.5×10^9/L;
   * PLT ≥ 80×10^9/L;
   * Hb ≥ 100g/L;
   * TBil ≤ 1.5 ULN;
   * ALB not lower than low limit of normal value;
   * BUN no more than high limit of normal value;
   * Cr ≤ 1.5 ULN high limit of normal value;
   * PT elongation ≤ 3 sec, APTT in normal value;
   * Fasting blood glucose ≤ 7.0mmol/L;
5. TSH in normal value;
6. AFP test result no more than high limit of normal value;
7. Take effective contraception for subject with child-bearing potential (including females and female partners of males);
8. Understand and sign ICF approved by EC;
9. Willing to comply with the study procedures and complete the study.

Exclusion Criteria:

1. Antibodies of HCV, HDV or HIV is positive;
2. ANA titer > 1:100;
3. Decompensated liver disease (such as gullet and pylorus varicose veins, hepatic encephalopathy);
4. Have the following illness or with severe disease inappropriate to participate in the study in the view of the investigator, in cardiovascular system: instable or significant cardiovascular illness such as angina pectoris, heart attack of myocardial infarction, congestive heart failure, severe hypertension, significant arrhythmia or abnormal ECG etc;

   * Respiratory system: bronchiectasia, bronchial asthma, chronic obstructive pulmonary disease, respiratory failure, etc;
   * Endocrine, metabolism diseases: diabetes mellitus, uncontrolled thyroid diseases, etc;
   * Others: autoimmune disorder, active tuberculosis, malignancies (e.g.: tumor), neuropathic, metal, acute or chronic pancreatitis illness history, etc.
5. Have used anti-HBV drug ( Interferon, Lamivudine, Adefovir Dipivoxil, Entecavir and Telbivudine ) and immunomodulator ( Thymic peptide, etc ) to the administration of study medication;
6. Have allergic diathesis or have suspected allergy to εPA-44;
7. Female in pregnancy, lactation or those who plan to pregnancy during the course of the study;
8. Have history of alcohol abuse (Alcohol consumption for more than 5 years, with daily consumption over 40g for males and over 20g for females) and known drug dependence;
9. Have history of organ transplantation (except corneal transplantation and hair transplantation);
10. Have participated in any other drug clinical investigations within 3 months;
11. Any other factors inappropriate for enroll in the study or study completion in the view of the investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 378 (Actual)
Dates: Start 2010-06 (Actual); Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: LanJuan Li, Ph.D., Principal Investigator — Zhejiang University
Locations (15):
- China (15):
  - The First Affiliated of Anhui Medical University, Hefei, Anhui
  - Beijing Youan Hosptial,Capital Medical University, Beijing, Beijing Municipality
  - The Third People's Hosptial of Shenzhen, Shenzhen, Guangdong
  - Renmin Hosptial of Wuhan University, Wuhan, Hubei
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - Xiangya Hospital Central South University, Changsha, Hunan
  - 81th Hospital of PLA, Nanjing, Jiangsu
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - The Second Hospital of Nanjing, Nanjing, Jiangsu
  - TangDu Hospital, XiAn, Shanxi
  - First Affiliated Hospital of Kunming Medical University, Kunming, Yunnan
  - The First Affiliated Hospital of Zhejiang University, Hangzhou, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang
  - 302 Militray Hosptial of China, Beijing
  - Southwest Hospital, Chongqing

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Therapeutic HBV Vaccine+Entecavir | Placebo+Entecavir
Started | 189 | 189
Completed | 172 | 176
Not Completed | 17 | 13
Not completed — Lost to Follow-up | 8 | 7
Not completed — Protocol Violation | 3 | 4
Not completed — Pregnancy | 0 | 1
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 5 | 1

BASELINE CHARACTERISTICS:
Population: Population analysis based on intention to treat
Groups:
- Total: Total of all reporting groups
Arm/Group | Therapeutic HBV Vaccine+Entecavir | Placebo+Entecavir | Total
Number analyzed (Participants) | 189 | 188 | 377
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.2 (9.52) | 28.3 (7.91) | 28.7 (8.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 46 | 87
  Male | 148 | 142 | 290
BMI [Mean (Standard Deviation); unit: kg/m^2] — Body Mass Index
  kg/m^2 | 21.61 (2.707) | 21.78 (3.014) | 21.7 (2.861)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With HBeAg Seroconversion at Week 48
Description: Primary endpoint data were summarised under "End of Study",using the last available post-baseline observation(Last Observation Carried Forward,LOCF)
Time Frame: 48 weeks
Population: Intention-To-Treat Population
Measure: Count of Participants; unit: Participants
Arm/Group | Therapeutic HBV Vaccine+Entecavir | Placebo+Entecavir
Number analyzed (Participants) | 189 | 188
Participants | 21 | 23

2. Secondary Outcome: Serological Response
Description: Serological response at every observation time: serological conversion rate of HBeAg, negative conversion rate of HBeAg, and change of HBeAg.
Time Frame: 96 weeks
Reporting Status: Not Posted

3. Secondary Outcome: Virological Response
Description: Virological response at every observation time: the proportion of patients with serum HBV DNA level reduction to undetectable level, decreased amount of serum HBV DNA compared with the baseline value, and HBV DNA load decrease 2 log scales or HBV DNA level <1.72×104 IU/ml.
Time Frame: 96 weeks
Reporting Status: Not Posted

4. Secondary Outcome: Biochemistry Response
Description: Biochemistry response at every observation time, mean the ALT level reduce to normal.
Time Frame: 96 weeks
Reporting Status: Not Posted

5. Secondary Outcome: Histological Response
Description: Histological response at week 72, mean histological score limited reduce 2 (reduced score 2-5), and no fiber deterioration compare with before treatment.
Time Frame: 72 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: After doing(0-96week)
Arm/Group | Therapeutic HBV Vaccine+Entecavir | Placebo+Entecavir
All-Cause Mortality (participants affected / at risk) | 0/189 | 0/189
Serious Adverse Events (participants affected / at risk) | 1/189 | 0/189
Other Adverse Events (participants affected / at risk) | 38/189 | 54/189
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Therapeutic HBV Vaccine+Entecavir (N=189) | Placebo+Entecavir (N=189)
Anaphylactic shock (Immune system disorders) | 1 (1) | 0 (0) — The subjects had no history of anaphylaxis prior to private prosecution, and anaphylactic shock occurred after the sixth injection of the drug, which was recovered after shock treatment
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Therapeutic HBV Vaccine+Entecavir (N=189) | Placebo+Entecavir (N=189)
upper respiratory infection (Infections and infestations) | 10 | 10
nasopharyngitis (Infections and infestations) | 21 | 24
Diarrhea (Gastrointestinal disorders) | 2 | 8
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 6
Dizziness (Nervous system disorders) | 4 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigators can't publish articles relevant to the study unless the sponsor permits.